CLINICAL TRIAL: NCT00598546
Title: Quality of Life Among Long-Term Survivors of Resected Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Coit, Daniel, MD / Pricipal Investigator, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 04-112
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Gastric Cancer
Keywords: Stomach; Gastric; Stomach Tumor; Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1
  Interventions: Behavioral: EORTC QLQ-C30, QLQ-STO22, and MSK-10

INTERVENTIONS:
Behavioral: EORTC QLQ-C30, QLQ-STO22, and MSK-10 — QLQ-C30 is the generic QOL tool for patients with cancer undergoing clinical trials.QLQ-STO22, containing 22 questions specific to gastric cancer, is currently the only standardized disease-specific questionnaire to measure the QOL of gastric cancer and must be used in conjunction with the QLQ-C30.MSK-10 consists of ten additional questions that were developed by surgeons on the GMT service to answer specific questions about outcomes related to proximal subtotal, distal subtotal, and total gastrectomies. These questions focus on eating capabilities, work status and major life changing events.

SUMMARY:
The purpose of this study is to find out how you feel about the quality of your life after having had surgery to remove your stomach tumor. Some patients continue to experience different problems after stomach surgery, even when the surgery was more than three years ago. The purpose of this study is to find out the specific things that may continue to affect patients' quality of life after a major operation.

DETAILED DESCRIPTION:
The purpose of this study is to measure the quality of life (QOL) of long-term survivors of resected gastric cancer. This cohort of long-term survivors will include patients who have no evidence of disease (NED) at least three years after having curative resection for gastric cancer. There are three main types of surgical procedures used to resect primary gastric cancer, which include proximal subtotal, distal subtotal, and total gastrectomy. Surgical management of gastric cancer at Memorial Sloan-Kettering Cancer Center (MSKCC) has shifted over the years to a greater use of proximal subtotal gastrectomies than in the past; however the effects on the QOL of these patients are unknown. In this study, we propose to use the European Organization for Research Treatment of Cancer (EORTC) two-part questionnaire QLQ-C30 and QLQ-STO22. This instrument has been shown to be a valid and reliable QOL instrument used to assess the quality of life of patients with gastric cancer.

We will measure multiple domains of QOL including, physical, role, cognitive, and emotional functions. An additional 10-item questionnaire (MSK-10) was designed by GMT service surgeons and will be administered in order to more specifically identify certain potential issues of QOL among gastric cancer survivors. These issues include eating capabilities, work status and major life changing events. Patients will be identified using the Gastric and Mixed Tumor (GMT) Service Gastric Cancer Database. The questionnaires will be conducted via telephone interview. Establishing these QOL measurements will help to provide valuable baseline data upon which to base future clinical trials of optimal surgical techniques.

OBJECTIVES AND SCIENTIFIC AIMS

* To establish health related QOL using the EORTC QLQ-C30 and QLQ-STO22 in gastric cancer patients who are alive and free of disease for three or more years after a proximal, distal, or total gastrectomy for gastric cancer.
* To compare the differences in QOL scores between the three different types of gastrectomy.
* To compare results using the EORTC QLQ-C30 with published norms established in the United States.
* To use the MSK-10 to assess the incidence and degree of certain areas of QOL that may affect gastric cancer survivors specifically.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age 18 or older
* Diagnosis of adenocarcinoma of the stomach
* Patient had curative surgical resection, including proximal, distal, or total gastrectomy
* Patient is at least three years NED
* Provide informed consent
* Fluent in English

Exclusion Criteria:

* Psychiatric or psychological abnormality precluding informed consent or ability to complete questionnaires
* Non-psychiatric disorder causing a lack of capacity to give consent or an inability to complete questionnaires (ie dementia, stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had curative resection at MSKCC for gastric cancer and are at least three years NED.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Instrument: EORTC QLQ-C30, QLQ-STO22, and MSK-10. The intent of this study is to assess QOL in long-term survivors of all surgical procedures performed for the treatment of gastric cancer. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Coit, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org